CLINICAL TRIAL: NCT01992432
Title: A Pilot Study of Structural and Functional Brain Magnetic Resonance Imaging Findings of Chemotherapy Toxicity in Older Women With Breast Cancer
Brief Title: Brain Functional MRI in Older Women With Breast Cancer (Brain fMRI-BC)
Acronym: Brain fMRI-BC
Status: Active, not recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 13278; 1R03AG045090 (NIH)
Record Dates: First submitted 2013-11-14; First posted 2013-11-25 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Brain magnetic resonance imaging; chemotherapy toxicity; older woman; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Single-group study: chemotherapy: Single-group study: chemotherapy

SUMMARY:
This study will use advanced MRI techniques to characterize the changes that occur to the structure and functionality of the brain in older breast cancer patients receiving adjuvant chemotherapy, and determine the relationship between the brain changes and severity of chemotherapy toxicity. Our results will be an early step towards identifying neuroimaging markers of aging, breast cancer and chemotherapy treatment, and will contribute to our understanding of the underlying pathophysiology of cognitive changes and chemotherapy toxicity in vulnerable, older adults with cancer. Furthermore, the work will lay the foundation for future, larger scale clinical studies of cognitive changes and chemotherapy toxicity in the aging cancer population.

DETAILED DESCRIPTION:
Breast cancer is the leading cancer diagnosed among woman in the US and is the second leading cause of cancer deaths. Adjuvant chemotherapy has been proven to decrease the risks of relapse and mortality from breast cancer. However, older adults are at increased risk for chemotherapy toxicity, including an increased risk of treatment-related mortality. At present, there is only preliminary evidence regarding which brain structures and functions are affected by chemotherapy and toxicity in breast cancer patients. However, this prior research did not specifically study older women. Thus, there is a need to establish a more sensitive test that has reproducible biomarkers, to identify the older breast cancer patients who are at higher risk for chemotherapy toxicity Our long term goal is to identify highly sensitive and reproducible brain MRI biomarkers that are associated with chemotherapy toxicity in aging cancer patients. Toward that goal, the objective of this study is to define the changes that occur on brain MRI and to determine the relationship between brain MRI changes and chemotherapy toxicity in older adults with breast cancer. We aim to 1) define structural and functional changes that occur on brain MRI of older women with breast cancer receiving adjuvant chemotherapy and; 2) determine the relationship between the severity of structural and functional changes on brain MRI and chemotherapy toxicity. We expect that the severity of structural and functional changes to the brain MRI in our patients will correlate with the severity of chemotherapy toxicity. The proposed study is significant because it focuses on the unknown relationship between brain MRI changes and chemotherapy toxicity in older women with breast cancer. It is innovative because it proposes advanced MRI techniques to study and identify the novel potential biomarkers for chemotherapy toxicity in older adults with breast cancer. It will have a positive impact by helping to clarify the underlying pathophysiology of cognitive decline caused by chemotherapy toxicity. The data generated from this pilot study will also help to serve as a foundation for future large scale studies of cognition and chemotherapy in older adults.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients with stage I-III breast cancers who are to receive adjuvant chemotherapy;
* 2) Able to understand English (the functional MRI task paradigms and neurocognitive testing are not validated in languages other than English);
* 3) Able to provide informed consent;
* 4) Patients age ≥ 65 and of any performance status.

Exclusion Criteria:

* 1) Patients with metastatic disease;
* 2) Patients with MRI exclusion criteria such as claustrophobia, cardiac pacemaker, and orbital metal implants.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Using a prospective longitudinal study design, 25 patients will be recruited for this study from the outpatient medical oncology practice at City of Hope Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Intensity of brain activation during functional brain MRI. | 2 years
  Prior to and after chemotherapy in older patients with breast cancer.

SECONDARY OUTCOMES:
NIH Tool box cognitive assessment. | 2 years
  Secondary measures include the changes in cognitive assessment measured by NIH Toolbox cognitive testing prior to and after chemotherapy.
Structural MRI brain parameters. | 2 years
  These secondary measures include gray matter density, fractional anisotropy (FA) and resting-state brain connectivity.
Chemotherapy toxicity. | 2 years
  Chemotherapy toxicity as a secondary outcome measure will be captured in a standardized manner using the NCI Common Toxicity Criteria for Adverse Events (v4.0) (NCI CT CAE version 4.0). Furthermore, we will determine the association of the brain MRI parameters for both structure and function with chemotherapy toxicity in older patients with breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Bihong T. Chen, MD., Ph.D, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - South Pasadena Cancer Center, South Pasadena, California

REFERENCES:
- [Background] Chen BT, Ghassaban K, Jin T, Patel SK, Ye N, Sun CL, Kim H, Rockne RC, Mark Haacke E, Root JC, Saykin AJ, Ahles TA, Holodny AI, Prakash N, Mortimer J, Waisman J, Yuan Y, Somlo G, Li D, Yang R, Tan H, Katheria V, Morrison R, Hurria A. Subcortical brain iron deposition and cognitive performance in older women with breast cancer receiving adjuvant chemotherapy: A pilot MRI study. Magn Reson Imaging. 2018 Dec;54:218-224. doi: 10.1016/j.mri.2018.07.016. Epub 2018 Aug 2. PMID 30076946
- [Derived] Chen BT, Ye N, Wong CW, Patel SK, Jin T, Sun CL, Rockne RC, Kim H, Root JC, Saykin AJ, Ahles TA, Holodny AI, Prakash N, Mortimer J, Sedrak MS, Waisman J, Yuan Y, Li D, Vazquez J, Katheria V, Dale W. Effects of chemotherapy on aging white matter microstructure: A longitudinal diffusion tensor imaging study. J Geriatr Oncol. 2020 Mar;11(2):290-296. doi: 10.1016/j.jgo.2019.09.016. Epub 2019 Nov 2. PMID 31685415
- [Derived] Chen BT, Jin T, Patel SK, Ye N, Sun CL, Ma H, Rockne RC, Root JC, Saykin AJ, Ahles TA, Holodny AI, Prakash N, Mortimer J, Waisman J, Yuan Y, Li D, Somlo G, Vazquez J, Levi A, Tan H, Yang R, Katheria V, Hurria A. Gray matter density reduction associated with adjuvant chemotherapy in older women with breast cancer. Breast Cancer Res Treat. 2018 Nov;172(2):363-370. doi: 10.1007/s10549-018-4911-y. Epub 2018 Aug 7. PMID 30088178
- [Derived] Chen BT, Sethi SK, Jin T, Patel SK, Ye N, Sun CL, Rockne RC, Haacke EM, Root JC, Saykin AJ, Ahles TA, Holodny AI, Prakash N, Mortimer J, Waisman J, Yuan Y, Somlo G, Li D, Yang R, Tan H, Katheria V, Morrison R, Hurria A. Assessing brain volume changes in older women with breast cancer receiving adjuvant chemotherapy: a brain magnetic resonance imaging pilot study. Breast Cancer Res. 2018 May 2;20(1):38. doi: 10.1186/s13058-018-0965-3. PMID 29720224